CLINICAL TRIAL: NCT01374451
Title: A Randomized, Open-label Phase II Multicenter Study Evaluating the Efficacy of Oral Everolimus Alone or in Combination With Pasireotide LAR i.m. in Advanced Progressive Pancreatic Neuroendocrine Tumors (PNET) - The COOPERATE-2 Study
Brief Title: Efficacy of Everolimus Alone or in Combination With Pasireotide LAR in Advanced PNET
Acronym: COOPERATE-2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped for not meeting the primary endpoint for PFS.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230I2201; 2010-023183-40 (EudraCT Number)
Record Dates: First submitted 2011-06-14; First posted 2011-06-16 (Estimated); Results first posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-10

CONDITIONS: Islet Cell Tumor
Keywords: Pancreatic; Neuroendocrine tumors; PNET; Pasireotide; Everolimus; Advanced progressive pancreatic neuroendocrine tumor
MeSH Terms: conditions — Adenoma, Islet Cell; Neuroendocrine Tumors; Neuroectodermal Tumors, Primitive | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paseriotide LAR + Everolimus (Experimental): everolimus 10 mg once daily po in combination with pasireotide LAR 60 mg every 28 days (q28d) im
  Interventions: Drug: Everolimus; Drug: Pasireotide LAR
- Everolimus (Experimental): everolimus 10 mg once daily po alone
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus was supplied as tablets of 5 mg strength, blister-packed under aluminum foil in units of 10 tablets
  Other Names: RAD001
Drug: Pasireotide LAR — Pasireotide LAR intra-muscular depot injections were supplied as a powder in vials containing 20 mg and 40 mg with ampoules containing 2 mL of vehicle (for reconstitution).
  Other Names: SOM230 LAR
  Arms: Paseriotide LAR + Everolimus

SUMMARY:
This study will estimate the treatment effect of everolimus in combination with pasireotide LAR relative to everolimus alone on progression-free survival (PFS) in patients with advanced progressive PNET.

A planned primary analysis was completed with data cut of 02-Apr-2014. The study did not meet its primary objective, which was based on progression-free survival (PFS) as per local radiology assessment and was prematurely terminated with the last patient last visit on 19-Feb-2015. However, it is important to note that the data did not reveal any new safety concerns. It was decided to stop the study and this decision was shared with the study sites on 31-Jul-2014.

ELIGIBILITY:
Inclusion Criteria:

* Advanced histologically confirmed well differentiated pancreatic neuroendocrine tumor
* Progressive disease within the last 12 months
* Measurable disease per RECIST Version 1.0 determined by multiphase MRI or triphasic CT

Exclusion Criteria:

* Patients currently requiring somatostatin analog treatment
* Prior therapy with mTOR inhibitors or pasireotide
* Patients with more than 2 prior systemic treatment regimens
* Previous cytotoxic chemotherapy, targeted therapy, somatostatin analogs, or biotherapy within the last 4 weeks

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (44):
- United States (4):
  - Dana Farber Cancer Institute SC-2, Boston, Massachusetts
  - Montefiore Medical Center MMC, The Bronx, New York
  - Oregon Health & Science University Knight Cancer Institute, Portland, Oregon
  - University of Texas/MD Anderson Cancer Center UT MD Anderson Cancer Ctr, Houston, Texas
- Argentina (2):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
- Australia (2):
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Herston, Queensland
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Haine-Saint-Paul
  - Novartis Investigative Site, Leuven
- Brazil (2):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Denmark (2):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen N
- France (5):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Villejuif
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, München
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- Italy (3):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
- Novartis Investigative Site, Fukuoka, Fukuoka, Japan
- Novartis Investigative Site, Rotterdam, Netherlands
- Novartis Investigative Site, Grafton, Auckland, New Zealand
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Madrid, Madrid
- Sweden (2):
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Uppsala
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Istanbul
- United Kingdom (3):
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Manchester

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paseriotide LAR + Everolimus | Everolimus
Started | 79 | 81
Completed | 78 | 81
Not Completed | 1 | 0
Not completed — Administrative problems | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) was defined according to the intention to treat principle. The FAS consisted of all randomized patients. Following the intention to treat principle patients were analyzed according to the treatment (and stratum) they were assigned to at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Paseriotide LAR + Everolimus | Everolimus | Total
Number analyzed (Participants) | 79 | 81 | 160
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.52 (11.978) | 58.22 (12.650) | 57.38 (12.314)
Gender [Count of Participants; unit: Participants]
  Female | 40 | 34 | 74
  Male | 39 | 47 | 86

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Per Local Radiological Review
Description: PFS per RECIST 1.0. (Response Evaluation Criteria in Solid Tumors). PFS was defined as the time from the date of randomization to the date of the first radiologically documented disease progression or death due to any cause.
Time Frame: Once 80 PFS events had occurred aproximately after 24 months
Population: The FAS consisted of all randomized patients. Following the intention to treat principle patients were analyzed according to the treatment (and stratum) they were assigned to at randomization.
  One patient in the everolimus + pasireotide LAR treatment arm was untreated due to administrative problems.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paseriotide LAR + Everolimus | Everolimus
Number analyzed (Participants) | 79 | 81
months | 16.82 [12.09 to 19.58] | 16.59 [11.07 to 19.48]
Statistical Analysis 1: Comparison: Paseriotide LAR + Everolimus vs Everolimus; Test type: Superiority or Other; p = 0.488, Log Rank; Hazard Ratio (HR) = 0.991, 95% CI 2-sided [0.636 to 1.543]

2. Secondary Outcome: Safety and Tolerability Profile of Everolimus Alone or in Combination With Pasireotide LAR
Description: Consisted of monitoring and recording the rate, type, severity, and causal relationship of adverse events (AEs) and serious AEs (SAEs) to treatment. The safety analysis was based mainly on the frequency of AEs or SAEs and on the number of laboratory values that fell outside of pre-determined range.
Time Frame: Once 80 PFS events had occurred
Population: Safety analysis population included all patients who received any study medication (i.e. at least 1 dose of the study drug in case of monotherapy or at least 1 dose of any 1 compound of the study treatment in case of a combination therapy) with a post-Baseline safety assessment.
  See Adverse Events (AE) section for all AEs collected.
Measure: Number; unit: Participants
Arm/Group | Paseriotide LAR + Everolimus | Everolimus
Number analyzed (Participants) | 78 | 81
Participants
  Deaths | 7 | 10
  Serious Adverse Events | 41 | 49
  Adverse Events | 78 | 81

3. Secondary Outcome: Objective Response Rate (ORR) as Per Radiology Review
Description: Objective response was determined by the local radiologist according to the RECIST Version 1.0. ORR is the percentage of patients with a best overall response of complete response (CR) or partial response (PR). This is also referred to as Overall response rate.
  CR: Disappearance of all nontarget lesions. PR: At least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the smallest sum of the longest diameter of all target lesions recorded at or after baseline.
Time Frame: Once 80 PFS events had occurred
Population: The FAS consisted of all randomized patients.1 patient in the everolimus + pasireotide LAR treatment arm was untreated due to administrative problems. The study was terminated because the study did not meet its primary objective so minimal efficacy data was obtained.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Paseriotide LAR + Everolimus | Everolimus
Number analyzed (Participants) | 79 | 81
Percentage of participants | 20.3 [12.0 to 30.8] | 6.2 [2.0 to 13.8]

4. Secondary Outcome: Duration of Response (DoR)
Description: 80 PFS are expected after approximately 24 months. Kaplan Meier was initially planned to be used to depict duration of response by treatment group and by stratum. Later based on the mode of action of everolimus and pasireotide and based on study experience, only a low number of objective responses per RECIST were expected. Therefore, protocol was amended to only list duration of response, and confirmed responses were flagged in the listing. Hence, statistical analyses were not planned and such data are not available for the following table.
Time Frame: Once 80 PFS events had occurred
Population: The FAS consisted of all randomized patients. Only a low number of objective responses per RECIST was expected. Therefore, protocol was amended to only list duration of response, and confirmed responses were flagged in the listing. Hence, statistical analyses were not planned and such data are not available for the following table.
Arm/Group | Paseriotide LAR + Everolimus | Everolimus
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival (OS) Using Kaplan Meier Method
Description: Overall survival was defined as the time from date of randomization/start of treatment to date of death due to any cause. If a patient is not known to have died, survival was to be censored at the date of last contact.
Time Frame: Once 80 PFS events had occurred
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Paseriotide LAR + Everolimus | Everolimus
Number analyzed (Participants) | 79 | 81
Percentage of participants
  6 months | 93.5 [85.0 to 97.2] | 93.7 [85.5 to 97.3]
  12 months | 85.5 [75.4 to 91.7] | 86.1 [76.2 to 92.0]
  18 months | 81.4 [70.6 to 88.5] | 75.5 [64.3 to 83.6]
  24 months | 77.0 [65.6 to 85.1] | 71.0 [59.3 to 79.9]

6. Secondary Outcome: PFS and the Predictive Probability of Success in Phase III
Description: 105 PFS events expected after approximately 36 months
Time Frame: Once 105 PFS events had occurred occurred
Population: Since the study was terminated because the study did not meet its primary objective which was based on PFS as per local radiology assessment, minimal efficacy data was obtained. Only 80 PFS events occurred before study was terminated so 105 PFS events was not reached to analyze this data.
Arm/Group | Paseriotide LAR + Everolimus | Everolimus
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Disease Control Rate (DCR) as Per Radiology Review
Description: Disease control rate is the percentage of patients with a best overall response of CR or PR or stable disease (SD) determined by the local radiologist according to the Response Evaluation Criteria In Solid Tumors Criteria (RECIST) Version 1.0. CR: Disappearance of all nontarget lesions. PR: At least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the smallest sum of the longest diameter of all target lesions recorded at or after baseline. SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease (PD). PD: Any progression ≤ 18 weeks after randomization (and not qualifying for CR, PR or stable disease SD.
Time Frame: Once 80 PFS events had occurred
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Paseriotide LAR + Everolimus | Everolimus
Number analyzed (Participants) | 79 | 81
Percentage of participants | 77.2 [66.4 to 85.9] | 82.7 [72.7 to 90.2]

8. Secondary Outcome: Summary of Pharmacokinetics (PK) for Everolimus for AUClast
Time Frame: Cycle 2 Day 1
Population: PK analysis set consisted of all patients who had at least 1 pasireotide LAR injection or 1 everolimus administration and 1 evaluable concentration data.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Paseriotide LAR + Everolimus | Everolimus
Number analyzed (Participants) | 5 | 8
ng*hr/mL | 511 (91.8) | 378 (123)

9. Secondary Outcome: Summary of Pharmacokinetics (PK) for Everolimus for CL/F
Time Frame: Cycle 2 Day 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Paseriotide LAR + Everolimus | Everolimus
Number analyzed (Participants) | 5 | 8
L/hr | 20.0 (3.21) | 29.0 (9.51)

10. Secondary Outcome: Summary of Pharmacokinetics (PK) for Everolimus for Cmax and Cmin
Time Frame: Cycle 2 Day 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paseriotide LAR + Everolimus | Everolimus
Number analyzed (Participants) | 6 | 9
ng/mL
  Cmax | 58.7 (25.9) | 60.2 (30.6)
  Cmin | 14.7 (4.81) | 7.67 (4.41)

11. Secondary Outcome: Summary of Pharmacokinetics (PK) for Everolimus for Tmax
Time Frame: Cycle 2 Day 1
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: hr
Arm/Group | Paseriotide LAR + Everolimus | Everolimus
Number analyzed (Participants) | 6 | 9
hr | 1.00 (4.81) [0.333 to 5.00] | 0.500 (4.41) [0.500 to 5.00]

12. Secondary Outcome: Summary of Pasireotide Concentrations Following Intramuscular Injection of Pasireotide LAR 60mg
Time Frame: Cycle 1 Day 21, Cycle 2 Day 29
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paseriotide LAR + Everolimus
Number analyzed (Participants) | 69
ng/mL
  Cycle 1 Day 21 (n:69) | 21.6 (13.1) [0.333 to 5.00]
  Cycle 2 Day 29 (n: 64) | 19.9 (12.1)

ADVERSE EVENTS:
Groups:
- Everolimus LAR + Pasireotide: everolimus 10 mg once daily po in combination with pasireotide LAR 60 mg every 28 days (q28d) im
Arm/Group | Everolimus LAR + Pasireotide | Everolimus
Serious Adverse Events (participants affected / at risk) | 41/78 | 49/81
Other Adverse Events (participants affected / at risk) | 77/78 | 80/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus LAR + Pasireotide (N=78) | Everolimus (N=81)
Anaemia (Blood and lymphatic system disorders) | 0 | 5
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Ocular icterus (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 5
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal oedema (Gastrointestinal disorders) | 0 | 1
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 | 0
Hernial eventration (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 3
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 0 | 2
Device occlusion (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 1
General physical health deterioration (General disorders) | 1 | 1
Localised oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Performance status decreased (General disorders) | 0 | 2
Pyrexia (General disorders) | 5 | 6
Cholangitis (Hepatobiliary disorders) | 2 | 3
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 2
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis aeromonas (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes simplex meningoencephalitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 4
Sinusitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood albumin decreased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 2
Blood glucose decreased (Investigations) | 1 | 0
Blood glucose fluctuation (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 1 | 1
C-reactive protein increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 3
Renal failure acute (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperaemia (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus LAR + Pasireotide (N=78) | Everolimus (N=81)
Anaemia (Blood and lymphatic system disorders) | 21 | 20
Leukopenia (Blood and lymphatic system disorders) | 3 | 7
Lymphopenia (Blood and lymphatic system disorders) | 4 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 9
Abdominal distension (Gastrointestinal disorders) | 7 | 8
Abdominal pain (Gastrointestinal disorders) | 22 | 29
Abdominal pain upper (Gastrointestinal disorders) | 10 | 15
Aphthous stomatitis (Gastrointestinal disorders) | 5 | 9
Constipation (Gastrointestinal disorders) | 11 | 18
Diarrhoea (Gastrointestinal disorders) | 49 | 43
Dysphagia (Gastrointestinal disorders) | 0 | 5
Flatulence (Gastrointestinal disorders) | 8 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 5
Mouth ulceration (Gastrointestinal disorders) | 4 | 6
Nausea (Gastrointestinal disorders) | 27 | 24
Steatorrhoea (Gastrointestinal disorders) | 9 | 2
Stomatitis (Gastrointestinal disorders) | 46 | 51
Toothache (Gastrointestinal disorders) | 3 | 5
Vomiting (Gastrointestinal disorders) | 22 | 15
Asthenia (General disorders) | 17 | 16
Fatigue (General disorders) | 21 | 27
Influenza like illness (General disorders) | 1 | 7
Non-cardiac chest pain (General disorders) | 1 | 6
Oedema peripheral (General disorders) | 26 | 31
Peripheral swelling (General disorders) | 4 | 4
Pyrexia (General disorders) | 15 | 21
Cystitis (Infections and infestations) | 7 | 3
Gastroenteritis (Infections and infestations) | 4 | 3
Influenza (Infections and infestations) | 5 | 6
Nasopharyngitis (Infections and infestations) | 12 | 10
Oral herpes (Infections and infestations) | 3 | 6
Pharyngitis (Infections and infestations) | 5 | 2
Pneumonia (Infections and infestations) | 1 | 5
Rhinitis (Infections and infestations) | 1 | 5
Upper respiratory tract infection (Infections and infestations) | 5 | 6
Urinary tract infection (Infections and infestations) | 4 | 5
Alanine aminotransferase increased (Investigations) | 5 | 4
Aspartate aminotransferase increased (Investigations) | 6 | 2
Blood alkaline phosphatase increased (Investigations) | 5 | 4
Blood lactate dehydrogenase increased (Investigations) | 4 | 1
Gamma-glutamyltransferase increased (Investigations) | 9 | 11
Glycosylated haemoglobin increased (Investigations) | 4 | 1
Haemoglobin decreased (Investigations) | 2 | 7
Weight decreased (Investigations) | 24 | 25
Decreased appetite (Metabolism and nutrition disorders) | 14 | 22
Diabetes mellitus (Metabolism and nutrition disorders) | 20 | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 16 | 15
Hyperglycaemia (Metabolism and nutrition disorders) | 56 | 23
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 10 | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 16 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 9 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 8
Dizziness (Nervous system disorders) | 4 | 5
Dysgeusia (Nervous system disorders) | 10 | 17
Headache (Nervous system disorders) | 17 | 26
Paraesthesia (Nervous system disorders) | 3 | 5
Anxiety (Psychiatric disorders) | 4 | 4
Insomnia (Psychiatric disorders) | 7 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 28
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 20
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 11
Acne (Skin and subcutaneous tissue disorders) | 1 | 7
Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 12 | 19
Nail disorder (Skin and subcutaneous tissue disorders) | 4 | 5
Onychoclasis (Skin and subcutaneous tissue disorders) | 5 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 18
Rash (Skin and subcutaneous tissue disorders) | 20 | 25
Hypertension (Vascular disorders) | 15 | 14

LIMITATIONS AND CAVEATS:
A planned primary analysis was completed with data cut of 02-Apr-2014. The study did not meet its primary objective, which was based on progression-free survival as per local radiology assessment and was prematurely terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.